CLINICAL TRIAL: NCT05778019
Title: Validation of Clavien-Madadi Classification for the Grading of Unexpected Events in Pediatric Surgery
Brief Title: Validating the Novel Classification for the Assessment and Grading of Unexpected Events in Pediatric Surgery: The Clavien-Madadi Classification
Acronym: ComPedS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Karolinska Institutet (Other); Helsinki University Central Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Ospedale dei Bambini Milano (Unknown); University of Leipzig (Other); Namik Kemal University School of Medicine, Tekirdag (Other)
Responsible Party: Sponsor
Other Study IDs: 9557_BO_K_2021_2
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Complication of Surgical Procedure
Keywords: Complications; Unexpected events; Severity Grading Systems; Classifications; Clavien-Madadi; Clavien-Dindo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Scenarios: No personal patient information is shared. The circulated case scenarios within the network will be constructed cases from the clinical practice, to serve representatively
  Interventions: Other: Case Scenarios of complications to be ranked / classified according to classifications (for the severity grading of events)

INTERVENTIONS:
Other: Case Scenarios of complications to be ranked / classified according to classifications (for the severity grading of events) — Test the feasibility, applicability and logic of a novel instrument for the grading of unexpected events in pediatric surgery (Clavien-Madadi classification) compared to the Clavien-Dindo classification for the grading of postoperative complications in general surgery
  Other Names: Comparison of the Clavien-Dindo and Clavien-Madadi classification

SUMMARY:
Despite appraisal of the Clavien-Dindo classification in the pediatric surgical literature, some criticize the transfer of the grading systems for adults in a pediatric cohort without modifications. In a recent study it has been shown that few items of the classification do not offer additional information in pediatric cohorts and organizational and management errors have been integrated, not being part of the initial proposal by Dindo et al.

In a group of pediatric and general surgeons, methodologists and statisticians of the ERNICA network the Clavien-Dindo classification has been modified for the application in pediatric surgery. The aim is to test and validate the novel Clavien-Madadi classification in a pediatric surgical cohort.

DETAILED DESCRIPTION:
Based on the protocol by Dindo et al. for the assessment of the international acceptability and reproducibility of the Clavien-Dindo classification, the aim is to circulate case scenarios (of complications/ unexpected events) within the ERNICA (European Reference Network for Rare Inherited Congenital Anomalies) network. Those case scenarios (15-20) should be graded by the respondents according to the Clavien-Dindo and Clavien-Madadi classification and preferences for future practice should be reported.

Milestones

1. All members of the working group send the PI´s 1-2 case scenarios with unexpected events in the management and treatment of neonates (preferably congenital diseases) and children for each grade of the Clavien-Madadi classification
2. All case scenarios will be circulated within the working group and will be ranked with a Likert scale (1 not accurate - 5 accurate) regarding the plausibility for an international survey
3. A final proposal of 15-20 case scenarios will be circulated within the working group
4. Circulating the case scenarios and the additional questionnaire via the ERNICA email distribution system and newsletter

ELIGIBILITY:
Inclusion Criteria:

* Case scenarios of unexpected events
* Case scenarios on neonatal surgery
* Case scenarios on congenital malformations
* Case scenarios with (re-)interventions
* Case scenarios with organ impairment
* Case scenarios with fatal result

Exclusion Criteria:

* Complex constructed case scenarios
* Case scenarios with adult patients
* Case scenarios with multiple events

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The constructed case scenarios will especially focus on congenital diseases, however, the spectrum of pediatric surgery (age: preterm infants to 17 years of age) will be included in the scenarios (if necessary)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Grading according to the Clavien-Madadi classification | Three months
  Grading of constructed case scenarios (by an international working group).
  Grading according to the Clavien-Madadi classification:
  Grade Ia - organizational and management errors Grade Ib - any deviation from the planned clinical course Grade II - pharmacological treatment Grade IIIa - Re-interventions (minimally-invasive) Grade IIIb - Re-interventions (laparotomy and / or thoracotomy) Grade IV - multiorgan dysfunction Grade V - death

SECONDARY OUTCOMES:
Grading according to the Clavien-Dindo classification | Three months
  Grading of constructed case scenarios (by an international working group)
  Grading according to the Clavien-Dindo classification:
  Grade I - any deviation from the planned postoperative course Grade II - pharmacological treatment Grade IIIa - Re-interventions not under general anesthesia Grade IIIb - Re-interventions under general anesthesia Grade IVa - single-organ dysfunction Grade IVb - multiorgan dysfunction Grade V - death
Comparison of Clavien-Madadi and Clavien-Dindo classification | Three months
  For each case scenario the respondents will have the option to select the superior classification (or specify no difference)

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
No individual participant data is necessary in our protocol. We will be focussing on constructed case scnearios, not including any specific patient data at all

REFERENCES:
- [Result] Sethi MV, Zimmer J, Ure B, Lacher M. Prospective assessment of complications on a daily basis is essential to determine morbidity and mortality in routine pediatric surgery. J Pediatr Surg. 2016 Apr;51(4):630-3. doi: 10.1016/j.jpedsurg.2015.10.052. Epub 2015 Oct 27. PMID 26628204
- [Result] Madadi-Sanjani O, Zoeller C, Kuebler JF, Hofmann AD, Dingemann J, Wiesner S, Brendel J, Ure BM. Severity grading of unexpected events in paediatric surgery: evaluation of five classification systems and the Comprehensive Complication Index (CCI(R)). BJS Open. 2021 Nov 9;5(6):zrab138. doi: 10.1093/bjsopen/zrab138. PMID 35022674
- [Result] Madadi-Sanjani O, Brendel J, Uecker M, Pfister ED, Baumann U, Ohlendorf J, Kuebler JF. Accumulation of Postoperative Unexpected Events Assessed by the Comprehensive Complication Index(R) as Prognostic Outcome Parameters for Kasai Procedure. Children (Basel). 2022 Oct 20;9(10):1590. doi: 10.3390/children9101590. PMID 36291526
- [Result] Madadi-Sanjani O, Brendel J, Kuebler JF, Ure BM. Definition, Documentation, and Classification of Complications in Pediatric Surgical Literature-A Plea for Standardization. Eur J Pediatr Surg. 2023 Apr;33(2):105-113. doi: 10.1055/s-0043-1760835. Epub 2023 Jan 31. PMID 36720251
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542